CLINICAL TRIAL: NCT02152254
Title: Randomized Study Evaluating Molecular Profiling and Targeted Agents in Metastatic Cancer: Initiative for Molecular Profiling and Advanced Cancer Therapy (IMPACT II)
Brief Title: Initiative for Molecular Profiling and Advanced Cancer Therapy (IMPACT II)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Tempus AI (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA12-1161; NCI-2016-00830 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA12-1161 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-05-21; First posted 2014-06-02 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Malignant Neoplasm; Recurrent Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Targeted Therapy (Active Comparator): Personalized treatment, targeted therapy against the alteration based on molecular profiling.
  Interventions: Drug: Targeted Therapy Based on Molecular Profiling
- Arm B: Standard-of-Care Therapy (Experimental): Standard-of-Care treatment not selected on basis of alteration analysis.
  Interventions: Drug: Standard-of-Care Therapy

INTERVENTIONS:
Drug: Targeted Therapy Based on Molecular Profiling — Molecular profiling results are used to assign targeted therapy. Patients receive targeted therapy by participating in a Phase I or a Phase II clinical trial. If a clinical trial is not available, and a commercially available targeted therapy exists (Food and Drug Administration [FDA]-approved for another indication), patients can receive the FDA-approved drug.
  Arms: Arm A: Targeted Therapy
Drug: Standard-of-Care Therapy — Standard-of-care treatment regimen will be left to the discretion of the treating physician.
  Arms: Arm B: Standard-of-Care Therapy

SUMMARY:
This randomized clinical trial studies how molecular profiling and targeted therapy work in treating patients with cancer that has spread to other places in the body compared to standard treatment. Information about genetic differences in a patient's tumor can be used to choose treatment that may target the tumor. It is not yet validated whether selecting treatment after studying the genetic changes that are associated with cancer in a patient's tumor is a better way to treat patients with metastatic cancer compared to therapy not based on studying the genetic changes that are associated with cancer.

DETAILED DESCRIPTION:
I. To determine whether patients treated with a matched targeted therapy selected on the basis of genomic alteration analysis of the tumor have longer progression-free survival (PFS) than those whose treatment is not selected on the basis of alteration analysis. Genomic analysis of tumor sample will be performed at the time of enrollment to identify tumor molecular alterations and to assign treatment for every individual patient.

OUTLINE: After completion of molecular profiling, patients who qualify for the trial will be offered randomization as previously. If they wish to be randomized, patients will be randomized to one of the two arms: matched targeted therapy (ARM I) or other therapy (ARM II). Patients who decline to be randomized will then be offered their choice of the two trial arms.

ARM I: Matched targeted therapy: Molecular profiling results are used to assign targeted therapy. Patients receive targeted therapy by participating in a Phase I or a Phase II clinical trial. If a clinical trial is not available, and a commercially available targeted therapy exists (Food and Drug Administration [FDA]-approved for another indication), patients can receive the FDA-approved drug.

ARM II: Other therapy: Patients receive standard of care therapy at the discretion of the treating physician.

Patients with tumor progression who achieve the primary study endpoint can cross over to the other treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic cancer
* Patients may have received unlimited lines of prior therapy
* Prior to randomization, patients with metastatic disease must have been treated with established standard-of-care therapy, or physicians have determined that such established therapy is not sufficiently efficacious, or patients have declined to receive standard-of-care therapy
* The patient has measurable disease
* The patient has Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* The patient has biopsy-accessible tumor; for patients who had no prior anticancer therapy and had surgical resection within a year and tumor tissue is immediately available, that tumor will be analyzed and no biopsy will be needed
* Absolute neutrophil count >= 1,000/ul
* Platelets >= 100,000/ul (unless these abnormalities are due to bone marrow involvement)
* Total bilirubin level <= 1.5 x the upper limit of normal (ULN), unless the patient has known Gilbert's disease
* Alanine aminotransferase (ALT)/ serum glutamic pyruvic transaminase levels (SGPT) =< 2.5 X ULN (unless the patient has liver metastases)
* Serum creatinine clearance >= 50 ml/min by the Cockcroft-Gault formula
* If the patient has brain metastasis, they must have been stable (treated and/or asymptomatic) and the patient must have been off steroids for at least 2 weeks
* The patient has provided signed informed consent
* Patients with a previous malignancy (other than the patients' known cancer) that were treated successfully and are disease-free for at least 3 years are allowed
* Patients with a history of basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix are eligible
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; childbearing potential will be defined as women who have had menses within the past 12 months and who have not had a tubal ligation, hysterectomy, or bilateral oophorectomy; should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately
* Male subjects must agree to use effective contraception or abstinence while on study and for 90 days after last dose of study drug

Exclusion Criteria:

* Patients who are randomized to the control arm must not receive therapy based on prior molecular profiling
* The patient has received chemotherapy, surgery, or radiotherapy (for therapeutic purposes) within 3 weeks of initiating study treatment (4 weeks for bevacizumab or investigational drugs) or the patient has not recovered (grade >= 2 from side effects of the previous therapy); patients who receive palliative radiation therapy can be treated immediately after completion of radiation therapy
* The patient has cardiac conditions as follows: uncontrolled hypertension (blood pressure [BP] > 160/100) despite optimal therapy, uncontrolled angina, ventricular arrhythmias, congestive heart failure (New York Heart Association class II or above), baseline left ventricular ejection fraction (LVEF) =< 50%, prior or current cardiomyopathy, atrial fibrillation with heart rate > 100 beats per minute (bpm), unstable ischemic heart disease (myocardial infarction [MI] within 6 months prior to starting treatment or angina requiring use of nitrates more than once weekly)
* The patient has peripheral neuropathy >= grade 2
* The patient is pregnant (confirmed by serum beta human chorionic gonadotropin [b-HCG], if applicable) or is breastfeeding
* The patient has concurrent severe and/or uncontrolled medical disease that could compromise participation in the study (i.e., uncontrolled diabetes, severe infection requiring active treatment, severe malnutrition, chronic severe liver or renal disease)
* The patient has refractory nausea and vomiting or chronic gastrointestinal diseases (e.g., inflammatory bowel disease) or has had significant bowel resection that would preclude adequate absorption (for oral therapy only)
* The patient is unable to swallow capsules and/or has a surgical or anatomical condition that precludes swallowing and absorbing oral medication on an ongoing basis (for oral therapy only)
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1362 (Estimated)
Dates: Start 2014-05-13 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of Progression-Free Survival (PFS) Between the Two Randomized Arms | Continuous Monitoring, expected range from 2 months to 3 years
  Progression-free survival (PFS) of patients treated with a targeted therapy selected on the basis of mutational analysis of the tumor compared with PFS of those whose treatment is not selected based on alteration analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia M Tsimberidou, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Vo HH, Fu S, Hong DS, Karp DD, Piha-Paul S, Subbiah V, Janku F, Naing A, Yap TA, Rodon J, Ajani JA, Cartwright C, Johnson A, Song IW, Beck J, Kahle M, Nogueras-Gonzalez GM, Miller V, Chao C, Vining DJ, Berry DA, Meric-Bernstam F, Tsimberidou AM. Challenges and opportunities associated with the MD Anderson IMPACT2 randomized study in precision oncology. NPJ Precis Oncol. 2022 Oct 27;6(1):78. doi: 10.1038/s41698-022-00317-0. PMID 36302890
- [Derived] Naqvi MF, Vo HH, Vining D, Tsimberidou AM. Prolonged response to treatment based on cell-free DNA analysis and molecular profiling in three patients with metastatic cancer: a case series. Ther Adv Med Oncol. 2021 Mar 24;13:17588359211001538. doi: 10.1177/17588359211001538. eCollection 2021. PMID 33995588
- [Derived] Aletaha D, Alasti F, Smolen JS. Disease activity states of the DAPSA, a psoriatic arthritis specific instrument, are valid against functional status and structural progression. Ann Rheum Dis. 2017 Feb;76(2):418-421. doi: 10.1136/annrheumdis-2016-209511. Epub 2016 Jul 25. PMID 27457512
- See also: MD Anderson Cancer Center — http://www.mdanderson.org